CLINICAL TRIAL: NCT03744156
Title: Impact of CBT for Insomnia on Pain Symptoms and Central Sensitization in Fibromyalgia
Brief Title: Sleep and Pain Interventions in Women With Fibromyalgia
Acronym: SPIN-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Florida (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Christina McCrae, Professor, Psychiatry, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011835; 1R01NR017168-01A1 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2018-11-16 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia; Insomnia; Chronic Widespread Pain
MeSH Terms: conditions — Fibromyalgia; Sleep Initiation and Maintenance Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Treatment-Insomnia (Experimental): Cognitive Behavioral Treatment-Insomnia. 8 Session treatment focusing on behavior and cognitions related to sleep and pain.
  Interventions: Behavioral: Cognitive Behavioral Treatment-Insomnia
- Sleep Hygiene Education (Experimental): Sleep Hygiene Education. 8 Session treatment focusing on sleep hygiene education.
  Interventions: Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment-Insomnia — 8 session Cognitive Behavioral Therapy for Insomnia. Individualized sessions with a therapist.
  Other Names: CBT-I
  Arms: Cognitive Behavioral Treatment-Insomnia
Behavioral: Sleep Hygiene Education — 8 Session Sleep Hygiene Education. Individualized sessions with a therapist.
  Other Names: SHE
  Arms: Sleep Hygiene Education

SUMMARY:
Insomnia affects 67-88% of chronic pain patients. SPIN II is a randomized controlled clinical trial that will compare the effects of two cognitive behavioral sleep treatments in women with fibromyalgia and insomnia. This trial will yield important information about the roles of sleep, arousal, and brain structure and function in the development and maintenance of chronic pain in women with fibromyalgia.

DETAILED DESCRIPTION:
This mechanistic trial will assess sleep, pain, arousal, and neural imagining outcomes at baseline, post-8 week behavioral treatment (CBT-I or SHE), as well as at 6 and 12 month followups. This information will provide novel information about the neural structures and functional networks associated with chronic pain, and their manipulation through a cognitive behavioral intervention to improve insomnia. Demonstration that a relatively brief intervention can reverse or resolve pain related maladaptive neural plasticity, and improve or resolve clinical pain symptoms would have immediate and far-reaching implications for millions of chronic pain sufferers as well as for the US healthcare system and economy.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18+ years of age
* willing to be randomized
* can read and understand English
* diagnosed with Fibromyalgia and insomnia
* no prescript or over the counter pain or sleep medicaments for 1+ month

Exclusion Criteria:

* unable to provide informed consent
* cognitive impairment
* sleep disorder other than insomnia (i.e., sleep apnea, periodic limb movement disorder
* bipolar or seizure disorder
* other major psychopathology (other than depression or anxiety)
* psychotropic or other medications that alter pain or sleep
* participation in non-pharmacological treatment (including CBT) for pain, sleep, or mood outside current trial
* internal metal objects or electrical devices
* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Self-Reported Bedtime, Wake time, Sleep Onset Latency, Wake After Sleep Onset, Sleep Quality on the Daily Diaries | baseline to follow-up (approximately 60 weeks)
  Participants will answer the following questions on the daily diaries:
  I napped for ____________ minutes yesterday. I napped ______ times yesterday. I napped in the ___morning ___afternoon ____evening (check all that apply) I went to bed last night at ____________ AM/PM. It took me ____________ minutes to fall asleep. I woke up ____________ times last night. I was awake for ____________ minutes in the middle of the night. My final wake up time was ____________ AM/PM. I got out of bed at ____________ AM/PM. I would rate my quality of sleep last night as ____________.
  1. very poor 2. poor 3. fair. 4 good 5. Excellent
Change in Insomnia Severity Index (ISI) | baseline to follow-up (approximately 60 weeks)
  The Insomnia Severity Index will be administered four times - baseline, post-treatment, and 6 and 12 month follow-up. Analysis will involve examining the trend of change in the ISI.
Change in Peripheral Arousal | baseline to follow-up (approximately 60 weeks)
  heart rate variability (as measured by Holter-Monitoring)
Change in Perceived Stress Scale | baseline to follow-up (approximately 60 weeks)
  measures how much self-reported stress participants experience (from 0-never to 4-very often) across various 10 situations. Higher total scores indicate greater perceived stress.
Change in Dysfunctional Beliefs and Attitudes about Sleep (DBAS) | baseline to follow-up (approximately 60 weeks)
  30-item self-report questionnaire designed to identify and assess various sleep/insomnia-related cognitions (e.g., beliefs, attitudes, expectations, appraisals, attributions).
Change in Pain Catastrophizing Scale | baseline to follow-up (approximately 60 weeks)
  The PCS instructions ask participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales with the end points (0) not at all and (4) all the time. The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness. Total score range from 0-52, with higher scores indicating greater pain catastrophizing.
Change in self-reported ratings of Pain Sensitivity and Pain Unpleasantness on Daily Diaries | baseline to follow-up (approximately 60 weeks)
  Participants will rate how much pain they experience and how unpleasant the pain is on a scale of 1 to 100 on the daily dairies. Analysis will involve examining the trend of changes in these ratings.
Neural Imaging: Structural/Functional MRI/Diffusion Weighted Imaging | baseline to follow-up (approximately 60 weeks)
  assessment of neural plasticity
Change in Bedtime, Wake time, Sleep Onset Latency, and Wake After Sleep Onset measured by Actigraphy | baseline to follow-up (approximately 60 weeks)
  Actiwatch-L (ACT-L; Mini Mitter, Inc.) will be used to obtain a behavioral measure of sleep outcome. ACT-L is a wristwatch-like device that provides long-term monitoring of ambient light exposure and gross motor activity in human subjects. The Actiware-Sleep software provides behavioral estimates for several sleep variables: (1) sleep onset latency-interval between bedtime and sleep start; (2) total sleep time-sum of all sleep epochs within the sleep period; (3) sleep efficiency percentage- ratio of total sleep time to total time spent in bed × 100; and (4) total wake time-sum of all wake epochs within the sleep period.
Change in Thermal Pain Response | baseline to follow-up (approximately 60 weeks)
  Participants will undergo quantitative sensory testing using a contact thermode applied to the volar surface of the forearm. The protocol that will assess both first pain (primarily A-delta function) and second pain (primarily C-fiber input). All thermal stimuli will be delivered using a computer-controlled Medoc Thermal Sensory Analyzer (TSA-2001, Ramat Yishai, Israel).
  Visual Analog Scale (VAS) ratings of 4 graded intensities (45, 47, 49, 51° C) of 5 second temperature stimuli will be obtained in the following fashion: Stimulus presentation will be timed such that no site is stimulated with less than a 3-minute interval to avoid sensitization of the site. Participants will rate 8 stimuli (2 at each intensity) using a VAS for pain intensity anchored at the right end by "the most intense pain imaginable." A second random sequence of 8 stimuli (2 at each intensity) will be rated by VAS for pain unpleasantness.

SECONDARY OUTCOMES:
Polysomnographically assessed sleep onset, wake time after sleep onset, sleep efficiency, number of awakenings, total sleep time, and sleep stage %. | baseline to follow-up (approximately 60 weeks)
  Ambulatory Polysomnography will be conducted four times at baseline, post-treatment, 6-month, and 12 month follow-up. This involves attachment of small electrodes and wires to the head and body.
Change in pain severity assessed by the McGill Pain Questionnaire | baseline to follow-up (approximately 60 weeks)
  The McGill Pain Questionnaire will be administered four times - baseline, post-treatment, 6 month and 12 month follow-up. Analysis will involve examining the trend of change in the scores in McGill Pain Questionnaire.
Change in pain-associated disability assessed by the Pain Disability Questionnaire | baseline to follow-up (approximately 60 weeks)
  The Pain Disability Questionnaire will be administered four times - baseline, post-treatment, 6 month follow-up and 12-month follow-up. Analysis will involve examining the trend of change in the scores in Pain Disability Questionnaire.
Change in Beck Depression Inventory-Second Edition | baseline to follow-up (approximately 60 weeks)
  This 21-item scale measures self-reported depressive symptoms. Total scores range from 0-63, with higher scores indicating greater maladjustment.
Change in State-Trait Anxiety Inventory-Form Y1 (STAI-YI) | baseline to follow-up (approximately 60 weeks)
  The STAI-Y1 contains 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Change in Pain Anxiety Symptoms Scale | baseline to follow-up (approximately 60 weeks)
  A 20 item self-report scale that measures the frequency (0-never, to 5-almost always) of anxiety across situations in which pain is experienced. Total scores range from 0 to 100 with higher scores indicating greater anxiety related to pain.
Change in Anxiety and Preoccupation about Sleep Questionnaire | baseline to follow-up (approximately 60 weeks)
  A 10-item scale that asks participants to rate the level of worry and/or anxiety during several situations regarding disturbed sleep. Participant rate the truthfulness of each statement according to their own experience (1-not true to 10-very true). Higher total scores indicate greater anxiety/preoccupation about sleep.
Activities of Daily Living (ADL) - Katz ADL Scale | baseline to post-treatment (approximately 12 weeks)
  A 6-item scale that measures the degree of independence on activities of daily living (1-independent; 0-dependent; activities include bathing, dressing, toileting, transferring, continence and feeding). Higher total scores indicate greater degree of independence on ADLs
Independent Activities of Daily Living (IADL) - Lawton IADL Scale | baseline to post-treatment (approximately 12 weeks)
  A 8-item scale that measures the degree of independence in performing instrumental activities of daily living (1-independent; 0-dependent; instrumental daily activities include ability to use telephone, shopping, food preparation, housekeeping, laundry, transportation, responsibility for own medications, and finances). Higher total scores indicate greater degree of independence on IADLs
Cognitive Failures Questionnaire | baseline to post-treatment (approximately 12 weeks)
  A 25-item scale measuring subjective cognition; caregivers rate on a scale of 0 (never) to 4 (very often) how often they experience cognitive mistakes and errors in daily tasks
Cognition - NIH Toolbox | baseline to post-treatment (approximately 12 weeks)
  A 20-minute computerized battery completed in a single setting on iPad (20 in. screen); domains tested include processing speed and attention, visuospatial ability and memory, verbal learning and memory, and executive functioning and working memory
Hair Sample | baseline to post-treatment (approximately 12 weeks)
  A sample of hair (cut, not extracted/no hair bulb) will be analyzed for the inflammatory and stress hormone cortisol
Saliva Sample | baseline to post-treatment (approximately 12 weeks)
  A sample of saliva will be analyzed to determine if the APOE-4 genetic marker is present.
Biomarkers - Neurodegeneration and Inflammation | baseline to post-treatment (approximately 12 weeks)
  Blood based biomarkers and hormones will be examined at each assessment period; biomarkers include CRP & IL-6, AβB42, AβB40 & total tau and phosphorylated-Tau at threonine181 & threonine217
Plasma-Based Hormones | baseline to post-treatment (approximately 12 weeks)
  Blood plasma analysis of three hormones including estradiol, testosterone, and cortisol
Global Cognition - Mini Mental Status Exam (MMSE) | baseline to follow-up (approximately 60 weeks)
  An 11-item questionnaire that provides a measure of global cognition. Participants are asked questions related to orientation to time/place, memory immediate/ delayed recall, attention and calculation, naming, repetition, comprehension, reading, writing, and drawing. Participants are scored 0-incorrect or 1- correct on each item. Total score is computed (out of 30), with higher total scores indicating better global cognitive function.
Global Cognition - Montreal Cognitive Assessment (MoCA) | baseline to post-treatment (approximately 12 weeks)
  A 30-item questionnaire that provides a measure of global cognition. Participants are asked questions related to visuospatial/executive functioning, naming, memory immediate/delayed recall, attention, language, abstraction, and orientation to time/place. Participants are scored 0-incorrect or 1-correct on each item. Total score is computed (out of 30), with higher total scores indicating better global cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Christina McCrae, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri- Department of Psychiatry, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCrae CS, Curtis AF, Craggs J, Deroche C, Sahota P, Siva C, Staud R, Robinson M. Protocol for the impact of CBT for insomnia on pain symptoms and central sensitisation in fibromyalgia: a randomised controlled trial. BMJ Open. 2020 Sep 15;10(9):e033760. doi: 10.1136/bmjopen-2019-033760. PMID 32933953